CLINICAL TRIAL: NCT04476628
Title: Prospective Double-Cohort Study: Comparing Efficacy of Budesonide Via Delayed Release vs Immediate Release After Administration in the Lying Head Back Position
Brief Title: Efficacy of Budesonide Via Delayed Release vs Immediate Release
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Due to COVID-19, we didn't start this study
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Assistant Clinical Professor, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H20-00842
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Budesonide; MAD; CRS; Head Position; Timing of Release
MeSH Terms: conditions — Disease | interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided to either start with 5MR or 1MR administration methods. They will undergo a 2 week "washout" period before starting their respective administration method. The first administration methods will be once daily for 8 weeks in duration. This is then followed by an additional "washout" period of 2 weeks. Finally, patients will switch to the other administration method for an additional treatment duration of daily application for 8 weeks. We will assess which administration method is more effective. Patients will be asked to administer budesonide daily with a minimum requirement of at least five days a week to ensure changes seen are related to the appropriate treatment arm. The "washout" period will involve standard of care daily non-medicated intranasal saline irrigation. Data will be collected at baseline, 2 weeks, 10 weeks, 12 weeks, and lastly 20 weeks follow-up visit.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Budesonide 5MR then 1MR (Other): All participants will administer budesonide daily via Mucosal Atomization Device (MAD) with a minimum requirement of at least five days a week for the duration of the study in this arm.
  1. st time period: Patients will undergo a 2 week "washout" period. The "washout" period will involve standard of care daily non-medicated intranasal saline irrigation.
  2. nd time period: 5MR administration method once daily for 8 weeks in duration.
  3. rd time period: Patients will undergo a 2 week "washout" period of daily. The "washout" period will involve standard of care daily non-medicated intranasal saline irrigation.
  4. th time period: 1MR administration method once daily for 8 weeks in duration.
  Interventions: Drug: Budesonide; Device: Mucosal Atomization Device; Device: NeilMed squeeze bottle for Impregnated Nasal Saline Irrigation
- Budesonide 1MR then 5MR (Other): All participants will administer budesonide daily via Mucosal Atomization Device (MAD) with a minimum requirement of at least five days a week for the duration of the study in this arm.
  1. st time period: Patients will undergo a 2 week "washout" period. The "washout" period will involve standard of care daily non-medicated intranasal saline irrigation.
  2. nd time period: 1MR administration method once daily for 8 weeks in duration.
  3. rd time period: Patients will undergo a 2 week "washout" period of daily. The "washout" period will involve standard of care daily non-medicated intranasal saline irrigation.
  4. th time period: 5MR administration method once daily for 8 weeks in duration.
  Interventions: Drug: Budesonide; Device: Mucosal Atomization Device; Device: NeilMed squeeze bottle for Impregnated Nasal Saline Irrigation

INTERVENTIONS:
Drug: Budesonide — Budesonide is a corticosteroid that is commonly used intranasally to treat CRS.
  Other Names: Pulmicort
Device: Mucosal Atomization Device — MAD is a device used as an addition to a syringe to atomize medication to increase area of distribution. It is used to administer budesonide within the nasal passages and sinuses to administer medication for CRS.
Device: NeilMed squeeze bottle for Impregnated Nasal Saline Irrigation — INSI is delivered using a NeilMed squeeze bottle. It is used to administer budesonide within the nasal passages and sinuses to administer medication for CRS.
  Other Names: INSI

SUMMARY:
The aim of this study is to compare the efficacy of intranasal budesonide administration with lying head back position and a 5 mins time to release of medication (5MR) compared to 1 min time to release (1MR) in chronic rhinosinusitis patients (CRS). Participants will be instructed to administer via mucosal automatization device (MAD) with either of the two treatment approaches daily for 5 to 7 days per week and 8 weeks total. This is a crossover study design so each participants will be placed in the other treatment approach for an additional 8 weeks of treatment. Moreover, there will be a "washout" of 2 weeks after baseline assessment and before the first treatment, as well as a second "washout" of 2 weeks between the two treatment approaches. The participants will also complete study related procedures such as endoscopic evaluation, cultures, and two questionnaires throughout the study period. The investigators hypothesize that Budesonide delivered to the sinuses with a 5 minute time to release of medication will be more effective at decreasing inflammation when compared to a 1 minute time to release of medication after administration.

DETAILED DESCRIPTION:
Objective

To compare the efficacy of 1 minute versus 5 minutes time to release of budesonide with lying head back position following administration via mucosal atomization device (MAD).

Hypothesis

Budesonide delivered to the sinuses with lying head back position and a 5 minute time to release (5MR) of medication will be more effective at decreasing inflammation both objectively and subjectively when compared to 1 minute time to release (1MR) of medication after administration.

Baseline and Follow-up Visits Evaluation:

The following information will be obtained from each participant

Baseline Demographic Data: Age, sex, smoking status, CRS subtype, pre-existing comorbidities, history of asthma, history of previous surgery, history of previous medications including oral and inhaled corticosteroids.

Clinical Data: Modified Lund-Kennedy (MLK) scores, sinonasal cultures, Sino-nasal Outcome Test-22 (SNOT-22), EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) scores, and culture.

Conduct of Study:

The proposed study is a single blind randomized, controlled crossover study at of 20 weeks in duration. Participants who have CRS and who meet the inclusion and exclusion criteria, will be invited to participate in this study.

Participants will undergo a 2 week "washout" period before starting their respective administration method. The first administration methods will be once daily for 8 weeks in duration. This is then followed by an additional "washout" period of 2 weeks. Finally, participants will switch to the other administration method for an additional treatment duration of daily application for 8 weeks. The goal is to assess which administration method is more effective. Participants will be asked to administer budesonide daily with a minimum requirement of at least five days a week to ensure changes seen are related to the appropriate treatment arm. The "washout" period will involve standard of care daily non-medicated intranasal saline irrigation. Data will be collected at baseline, 2 weeks, 10 weeks, 12 weeks, and lastly 20 weeks follow-up visit. SNOT-22 questionnaires, EQ-5D-5L questionnaires, endoscopic evaluation, and Modified Lund Kennedy Scores will each be completed at baseline and then again at 2 weeks, 10 weeks, 12 weeks, and 20 weeks.

Upon enrolment in the study, participants will be randomly divided to either start with 5MR or 1MR administration methods through 1:1 block randomization. In addition, demographic data and clinical data will be obtained by the investigators.

Management of Patient Care:

The clinical care remains the same for participants participating in this study; however, there is a possibility that some participants will experience an increased frequency of visits to the clinic with some being spaced 2 weeks apart. The increased appointments are required to effectively transition each participants into the different treatment types and also to acquire additional outcome measures. This will be clearly explained to each participant to ensure that they are aware of the additional appointments compared to standard of care. Otherwise, there are no additional risks imposed on the study participants. Participants have the right to withdraw from the study at any time. Participants who meet any of the exclusion criteria that were not noted at the beginning of the study will be removed from this study and the physician will discuss the future management options with the participant.

Sample Size:

A recruitment goal of 60 participants (30 participants per study arm) is expected to demonstrate an effect for the study. To account for a drop-out rate of 25% the investigators plan to recruit 40 participants in each arm.

The washout periods included in the crossover study design will allow for more control in regards to reducing confounding variables. In particular, this allows participants to start at a similar baseline by using the same standard of treatment with Budesonide for the 2 weeks of washout before going into the 5MR or 1MR treatments.

Analysis:

Descriptive statistics will be used to analyze the baseline characteristic data and the data from the administered surveys and objective findings of cultures and MLK scores. In addition, rigorous statistical analysis will be conducted on the Likert scale-based SNOT-22 and EQ-5D-5L surveys. These analyses will include paired t tests with repeated measured ANOVA for validation and confidence intervals.

Safety Monitoring:

Participants who experience signs and symptoms of budesonide reaction will be noted and the code will be broken so that a discussion can occur between the research supervisor and the participants regarding the use.

All expected and unexpected adverse events will be recorded and graded by the research supervisor. Stable chronic conditions, which are present prior to the clinical trial entry and do not worsen, are not considered adverse events and will be accounted for in the participant's medical history.

During each participant visit, the research supervisor will ask appropriate questions and perform a physical exam to elicit any adverse events. The research supervisor will also review any relevant clinical data and laboratory investigations with the partcicpant. All reportable adverse events will be recorded on appropriate case report form. The research supervisor will also write the stop date, the severity of the AE and his judgment of the AE's relationship to the study.

A Serious Adverse Event (SAE) is defined as an AE meeting one of the following:

Death occurring between Day 0 and 182 days (6 months) of the study. Life Threatening Event (defined as a participant at immediate risk of death at the time of the event) In-participant hospitalization or prolongation of existing hospitalization between Day 0 and 42 of the study.

Results in a persistent or significant disability/incapacity In the event of SAE, the research supervisor will discuss with the partcipant (or next of kin) whether there is a relationship between the study and the SAE. If there is a relationship, the PI will be responsible for coordinating care for the participant until the SAE has been addressed.

Pregnancy During the Trial Participants will be responsible for determining if they are pregnant or become pregnant during the study. If participants notify the PI they are pregnant, they will be removed from the study and the medical management options will be discussed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 19 years and above
2. Patients with chronic or recurrent sinusitis (as defined by the American Academy of Otolaryngology) with or without nasal polyposis or allergic fungal rhinosinusitis.
3. Patients currently on budesonide or being prescribed budesonide for the first time
4. Minimum Modified Lund Kennedy score of 2.

Exclusion Criteria:

1. Individuals unable to understand the purpose, methods and conduct of this study
2. Patients unwilling to provide informed consent
3. Are immuno-compromised, and have impairment in mucociliary function (e.g., cystic fibrosis, Kartagener syndrome)
4. Have autoimmune diseases affecting the upper airway (eg Systemic lupus erythematosus, Sjögren's syndrome, systemic sclerosis etc)
5. Have sinonasal tumors
6. Patients with a history of pituitary disease
7. Patients with a known hypersensitivity to cortisol, corticotropin, or cosyntropin
8. Recent use of systemic corticosteroids such as prednisone (within last 3 months)
9. Patients who are pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Lund Kennedy Score | baseline and 20 weeks
  This score is based on the endoscopic assessment of polyps, edema, and discharge and are each given score 0-2. It is out of a total score of 12 with higher scores indicating a worse outcome.
Change in Sinonasal-Outcomes Test-22 (SNOT-22) Score | baseline and 20 weeks
  This is a standard of care baseline Sinonasal Outcome Test form that includes 22 questions about symptoms and social/emotional consequences of your nasal disorder. You will be asked to rate your problems as they have been over the past two weeks. An example of the questions is:
  * Need to blow nose
  * Sneezing It is out of a total of 110 and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) Score | baseline and 20 weeks
  This is a questionnaire that asks six multiple-choice questions about your mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and overall health. It is out of a total score of 100 and higher scores mean a worse outcome.
Change in sinus culture results | baseline and 20 weeks
  A swab will be taken from your nose to see if there are any bacteria or fungi present.

CONTACTS AND LOCATIONS:
Overall Officials: Amin JAver, MD, Principal Investigator — The University of British Columbia and St. Paul's Sinus Centre

IPD SHARING:
Plan to Share IPD: No
We will publish final outcomes as scientific paper.